CLINICAL TRIAL: NCT00746187
Title: An Open, Randomized Study to Compare Two Dental Implant Systems With Regard to Changes in Marginal Bone Level.
Brief Title: Study to Compare Marginal Bone Loss Around Implants From Two Dental Implant Systems.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-MIC-0003
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASTRA TECH Implant System; Fixture ST (Experimental): Ø 4.5 cm in lengths 9-13 mm
  Interventions: Device: ASTRA TECH Implant System; Fixture ST: Ø 4.5 cm in lengths of 9, 11 and 13 mm.
- Biomet 3i; Osseotite® Implants (Experimental): Ø 4.0 cm in lengths 8.5-13 mm
  Interventions: Device: 3i Osseotite® implant: Ø 4.0 in lengths of 8.5, 10, 11.5 and 13 mm

INTERVENTIONS:
Device: ASTRA TECH Implant System; Fixture ST: Ø 4.5 cm in lengths of 9, 11 and 13 mm.
  Arms: ASTRA TECH Implant System; Fixture ST
Device: 3i Osseotite® implant: Ø 4.0 in lengths of 8.5, 10, 11.5 and 13 mm
  Arms: Biomet 3i; Osseotite® Implants

SUMMARY:
The purpose of this study is to compare marginal bone level changes between ASTRA TECH Implant System; Fixture ST and Biomet 3i; Osseotite® Implants. Subjects with partial edentulism in the posterior maxilla and/or mandible will be included and a one-stage surgical protocol will be used. Implants will be loaded within 15 weeks from installation. The subjects will be followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Age 18 - 75 years
* Partial edentulism, Kennedy class I or II, last natural tooth must be cuspid or first bicuspid
* Edentulous in the area/s if implant placement for more than 2 months

Exclusion Criteria:

* Untreated caries and/or periodontal disease of residual dentition
* Need for pre-surgical bone or soft tissue augmentation in the planned implant area/s.
* Absence of occlusal stability in centric occlusion
* Any systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Pregnancy
* Present alcohol or drug abuse
* Tobacco smoking during the last 6 months
* Unable or unwilling to return for follow-up visits for a period of 3 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Tarnow, D.D.S. Prof., Principal Investigator — Dept. of Implant Dentistry, New York University (to March 2011); Stuart Froum, Dr, Principal Investigator — Dept. of Implant Dentistry, New York University (from March 2011)
Locations (2):
- United States (2):
  - Dept. of Implant Dentistry, New York University, New York, New York
  - Dept. of Prosthodontics, School of Dentistry, University of North Carolina, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- ASTRA TECH Implant System; Fixture ST: Ø 4.5 cm in lengths 9-13 mm
  ASTRA TECH Implant System; Fixture ST: Ø 4.5 cm in lengths of 9, 11 and 13 mm.
- Biomet 3i; Osseotite® Implants: Ø 4.0 cm in lengths 8.5-13 mm
  3i Osseotite® implant: Ø 4.0 in lengths of 8.5, 10, 11.5 and 13 mm
Period: Overall Study
Arm/Group | ASTRA TECH Implant System; Fixture ST | Biomet 3i; Osseotite® Implants
Started | 18 | 18
Completed | 15 | 16
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASTRA TECH Implant System; Fixture ST | Biomet 3i; Osseotite® Implants | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12) | 51 (11) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Level Changes
Description: Marginal bone adaptation was expressed as the distance from the implant reference point to the most coronal bone-to-implant contact on the mesial and distal side of the implant. Bone adaptation in millimeters at the 3-year follow-up visit were compared to values obtained at Implant placement (baseline). Positive value indicates bone gain and negative value bone loss.
Time Frame: 3 years after implant placement (baseline)
Population: Per protocol analysis presented and this includes 86 implants in 36 patients. At 3-year follow-up, 74 implants in 31 patients were still in the study and thus evaluable for the analysis.
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | ASTRA TECH Implant System; Fixture ST | Biomet 3i; Osseotite® Implants
Number analyzed (Participants) | 15 | 16
Number analyzed (Implants) | 36 | 38
millimeter | -0.25 (0.60) | -0.50 (0.93)

ADVERSE EVENTS:
Arm/Group | ASTRA TECH Implant System; Fixture ST | Biomet 3i; Osseotite® Implants
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ASTRA TECH Implant System; Fixture ST (N=18) | Biomet 3i; Osseotite® Implants (N=18)
Advanced breast cancer (Reproductive system and breast disorders) | 0 | 1
Prostate cancer (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less